CLINICAL TRIAL: NCT03634254
Title: Satisfaction Level of Communication Quality: a Survey for Primary Caregivers of AAC Users in New Taipei City
Brief Title: Satisfaction Level of Communication Quality
Acronym: slc
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201806068RINC
Record Dates: First submitted 2018-08-09; First posted 2018-08-16 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Complex Communication Needs
Keywords: AAC; Satisfaction level of communication quality

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- primary caregivers of AAC users in New Taipei City: Satisfaction level of communication quality
  Interventions: Other: Satisfaction survey of communication quality:

INTERVENTIONS:
Other: Satisfaction survey of communication quality: — a conversation from phone call to survey primary caregivers of AAC users in New Taipei City who think the users communication quality

SUMMARY:
This study mainly explores the actual situation of AAC users in New Taipei City in their daily life after applying for social security subsidies, and the satisfaction of the main caregivers to AAC actually helping case communication. In summary, the main purposes of this study are as follows:

1. Discuss the communication satisfaction of the main caregivers to AAC users.
2. Explore the barriers to AAC users applying AAC.

DETAILED DESCRIPTION:
This study was based on cross-sectional research, questionnaire survey, and the evaluation of the questionnaires by experts. The research tool part of the research and development reference to the domestic and foreign literature and questionnaires, developed a self-made questionnaire "communication quality satisfaction questionnaire", with continuous use and no continuous use of the auxiliary communication system as the self-variation in the study, in order to separately discuss the main caregiver Communication satisfaction of AAC users in different situations and activities in daily life, as well as obstacles in application

ELIGIBILITY:
Inclusion Criteria:

1. Apply for the communication from the New North City Access Center to identify the primary caregiver of the AAC users who have approved and purchased the AAC users.
2. The primary caregiver has normal communication skills and is interviewed by telephone.

Exclusion Criteria:

who may not participate in this study if you have any of the following conditions:

1. The main caregiver is unable to conduct telephone interviews due to physiological conditions (listening, deaf-mute)

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: primary caregivers of AAC users in New Taipei City
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-08-09 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-10-30 (Estimated)

PRIMARY OUTCOMES:
Satisfaction of communication quality | 1 times conversation from phone call about 15 mints
  a MEASURE Likert scalefor understand what satisfaction of communication quality about primary caregivers of AAC users in New Taipei City

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No